CLINICAL TRIAL: NCT00600899
Title: Use of Home Pumps for Analgesia After Ambulatory Foot Surgery - Comparison of Two Infusion Rates - a Randomized, Double-Blind Study
Brief Title: Home Infusors for Analgesia After Foot Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Dusanka Zaric, Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT2007-005180-10; 9445-DZ
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Hallux Valgus
Keywords: Postoperative pain treatment
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Group A patients will receive perisciatic continuous infusion of ropivacaine 2 mg/ml through an elastomeric pump (Baxter, Deerfield, IL, USA)) 8 ml/h (reservoir of 500 ml)as postoperative analgesia.
  Interventions: Procedure: elastomeric pump with reservoir of 500 ml, infusion rate of 8 ml/h
- B (Active Comparator): Group B patients will receive standard treatment: continuous perisciatic infusion of 2 mg/ml ropivacaine 5 ml/t (Baxter infusor with 275 ml reservoir)
  Interventions: Procedure: elastomeric pump with reservoir of 275 ml, infusion rate of 5 ml/h

INTERVENTIONS:
Procedure: elastomeric pump with reservoir of 500 ml, infusion rate of 8 ml/h — Continuous perisciatic infusion of ropivacaine 2mg/ml (Baxter infusor with 500 ml reservoir and infusion rate of 8 ml/h)
  Arms: A
Procedure: elastomeric pump with reservoir of 275 ml, infusion rate of 5 ml/h — Continuous perisciatic infusion of ropivacaine 2mg/ml (Baxter infusor with 275 ml reservoir and infusion rate of 5ml/h)
  Arms: B

SUMMARY:
The purpose of this double blind, randomized study is to evaluate which rate and duration of infusion can be recommended for continuous perisciatic infusion of ropivacaine 2 mg/ml for analgesia after ambulatory foot surgery.

DETAILED DESCRIPTION:
Protocol title:

Use of home pumps for analgesia after ambulatory foot surgery - comparison of two infusion rates SUMMARY in English

THE PURPOSE:

The purpose of this double blind, randomized study is to evaluate which rate and duration of infusion can be recommended for continuous perisciatic infusion of ropivacaine 2 mg/ml for analgesia after ambulatory foot surgery.

BACKGROUND:

In the previous study (1) we showed that the continuous perisciatic infusion of 2 mg/ml ropivacaine 5 ml/h for 55 hours provided better analgesia than placebo after ambulatory foot surgery. Similar results are reported by Singelyn (2), Ilfeld (3) and White (4). But, different pumps with different basal infusion rates were used in these studies. Singelyn used infusion rate of 7 ml/h for 48 hours, while Ilfeld used mechanical pump with adjustable infusion rate, starting with 8 ml/h and patient controlled analgesia (PCA) 2 ml/20 minutes for 2 postoperative days. In our and White's studies elastomeric pumps with reservoir of 500 ml and infusion rate of 5 ml/h were used in 55 hours. Capdevila (5) has shown that the patients prefer elastomeric pumps because they cause fewer problems. That is why it will be our choice as well.

The analgesic efficacy in our study was good as the patients in the treatment group had less pain and fewer sleep disturbances than in the placebo group. The question is whether higher infusion rate and longer duration would have an even better effect.

The aim of this study is to compare (in a double blind manner) two different regimens for continuous perisciatic nerve infusion of ropivacaine 2 mg/ml after ambulatory foot surgery:

1. elastomeric pump with reservoir of 275 ml, infusion rate of 5 ml/h (duration 55 hours) and
2. elastomeric pump with reservoir of 500 ml, infusion rate of 8 ml/h (duration 62 hours).

Design:

A randomized, double blind study with 40 ambulatory patients who will undergo foot or ankle surgery. These patients will be randomized to receive either regimen 1. (5 ml/h for 55 hours) or regimen 2. (8 ml/h for 62 hours). The randomization procedure: sequentially numbered, sealed, opaque envelopes that contain computer produced random numbers for treatment allocation. Blinding procedures: pre-numbered identical containers marked with "Test drug", date of production and infusion start/end will be provided by the registered nurse (SK). The patient and the acute pain nurse (EB), who will evaluate the effect of these two treatments, will be blinded.

On each of the 3 postoperative days the patients will be contacted by phone by the acute pain nurse and a standard questionnaire will be completed.

The primary effect variable is worst pain on the first postoperative day evaluated as VAS score.

ELIGIBILITY:
Inclusion Criteria:

* All ambulatory patients (ASA 1-3) scheduled for foot and ankle surgery in spinal or general anesthesia that are willing to participate in the study after informed consent will be taken into consideration.
* Age span: 19 -80 years.
* When fertile females are included, we will make sure that they receive anticonceptive treatment.

Exclusion Criteria:

* Contraindications for sciatic catheter placement and allergy to local anesthetics.
* The patients with chronic pain receiving opioids, pregnant patients, those with rheumatoid arthritis, lever or heart disease.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
worst pain | first postoperative day

SECONDARY OUTCOMES:
Average pain | 1st, 2nd and 3rd postoperative days
Opioid consumption | first, second and third postoperative days
Side effects | 1st, 2nd and 3rd postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Dusanka Zaric, MD pHd, Principal Investigator — Ndr. Fasanvej 57 2000 Frederiksberg
Locations (1):
- Frederiksberg Hospital, Frederiksberg, Denmark

REFERENCES:
- [Background] Zaric D, Boysen K, Christiansen J, Haastrup U, Kofoed H, Rawal N. Continuous popliteal sciatic nerve block for outpatient foot surgery--a randomized, controlled trial. Acta Anaesthesiol Scand. 2004 Mar;48(3):337-41. doi: 10.1111/j.0001-5172.2004.0327.x. PMID 14982567